CLINICAL TRIAL: NCT06997549
Title: Retrospective Analyses of the Greenbrook Database Evaluating Mental Health Treatments
Status: Recruiting | Type: Observational
Sponsor: Neuronetics (Other)
Responsible Party: Sponsor
Other Study IDs: 11-10002-000
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Depression; OCD; Anxiety Depression
MeSH Terms: conditions — Depression | interventions — Esketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Patients treated with NeuroStar TMS — non-invasive brain stimulation device
  Other Names: TMS
Drug: Patients treated with Esketamine — nasal spray for treating depression
  Other Names: spravato

SUMMARY:
The study involves multiple retrospective analyses to understand the utilization of mental health treatments provided at Greenbrook and their effectiveness

DETAILED DESCRIPTION:
this is a retrospective data analysis study that will utilize the already collected data as clinical care and will help understand the utilization and efficacy of various treatment options available for various mental heath conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female reported in database and not an invalid entry
* Age reported and not an invalid entry
* Treatment date in 2011 or later.

Exclusion Criteria:

• Incomplete information on treatment parameters

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who received mental health treatment at a Greenbrook Center and the data is available in their database.
Sampling Method: Probability Sample
Enrollment: 12000 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
change in clinical outcome scores from baseline to post treatment | 8 weeks
  real-world efficacy of NeuroStar TMS as compared to Esketamine in reducing patients' symptoms, reduction in clinical assessment score like PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Cole, PhD, Study Director — Neuronetics
Locations (1):
- Neuronetics, Malvern, Pennsylvania, United States